CLINICAL TRIAL: NCT04885192
Title: Implementation and Evaluation of a Virtually-Delivered, Stepped-Care Mental Health Treatment Program for Patients With Chronic Pain During COVID-19
Brief Title: Implementation and Evaluation of a Stepped-Care Mental Health Treatment Program for Patients With Chronic Pain
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Research Manager, University Health Network, Toronto
Other Study IDs: 20-6290
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
Keywords: Psychological Treatment; Stepped-Care; Virtual Care
MeSH Terms: conditions — Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stepped-Care Model — Step 0: Screening via Manage My Pain (MMP) App. Patients using MMP will be prompted to complete questionnaires on pain catastrophizing, depressive symptoms, anxiety, suicide risk and opioid risk. Those scoring above clinical risk cut-offs will be referred to Step 1.
  Step 1: Acceptance and Commitment Therapy (ACT) Workshop. Patients will be offered a virtual ACT workshop focusing on practical coping skills for dealing with pain, emotional dysregulation, and disability, while maximizing functioning and quality of life with chronic pain. Thirty days later, patients will be prompted to complete all questionnaires through MMP again; those who score above clinical risk cut-offs will be referred to Step 2.
  Step 2: Dialectic Behavior Therapy (DBT) group. A 6-week DBT-based skills group will cover topics such as self-compassion, radical acceptance, distress tolerance, and mindfulness, among others. Thirty days later, patients will be prompted to complete questionnaires through MMP.
  Other Names: Psychological screening; Acceptance and Commitment Therapy; Dialectic Behavior Therapy

SUMMARY:
Chronic pain affects nearly 20% of Canadians, and sixty percent or more of individuals with chronic pain are also struggling with mental health or substance use disorders (referred to as complex chronic pain, or CCP, patients). This is a major concern in the best of times and has become an emergency during the COVID-19 pandemic. Now individuals suffering from chronic pain are faced with the additional challenges of quarantine, including the stress of isolation, delays in much needed medical care, and anxiety of possible infection to self or loved ones. Prior to COVID-19, psychologists at The Transitional Pain Service and the GoodHope Ehlers-Danlos Syndrome Clinic at Toronto General Hospital have adapted gold standard treatments for mental health and substance use for the unique needs of individuals with CCP. The investigators propose to develop these treatments into a virtual intervention that will meet the needs of patients during and after the COVID-19 pandemic. The investigators will use a mobile health application (called Manage My Pain or MMP) already in use by our patients to identify patients with CCP currently struggling with mental health issues or at risk of opioid misuse. Patients identified at risk will be offered a single-session Acceptance and Commitment Therapy workshop and then reassessed one month after the workshop. Patients still reporting high levels of emotional distress or substance use risk at that time will be offered a six-week Dialectic Behavior Therapy-informed group and will be reassessed one month after conclusion of the group. The investigators propose to conduct prospective data collection during the implementation of this program to facilitate 1) evaluation of the impact of stepped-care program components on mental health and substance use concerns, 2) examination of current rates mental health and substance use concerns in patients, and 3) examination of uptake for virtual mental health care amongst patients with chronic pain.

DETAILED DESCRIPTION:
Mood and anxiety disorders are 2 to 7 times more prevalent in patients with chronic pain, and comorbid chronic pain and psychiatric conditions results in poorer prognosis.(1) Patients with chronic pain struggle to gain control of their disease and a significant proportion of these patients are on high dose opioids (i.e. greater than 90 mg of morphine equivalents/day).(2) Treatment of chronic pain in the context of mental distress/psychological comorbidity and/or opioid use is complex and the investigators have therefore adopted the term 'complex chronic pain' (CCP) to identify the unique needs of these patients.

Due to public health measures to control the spread of COVID-19, pain clinics across the country have ceased or severely restricted in-person visits,(3) which significantly impacts care of the 15-19% of Canadians who struggle with chronic pain.(4) Thus, chronic pain patients have lost resources that were their mainstay of stability such as routine physiotherapy and psychotherapy. Moreover, additional stresses related to social isolation, delay of medical procedures that reduce symptoms and improve quality of life, and anxiety regarding possible COVID-19 infection or impact from actual infection on self or loved ones further impact mental health. This is reflected in a recent survey of multidisciplinary Canadian pain clinics where increased pain, stress, and opioid use has been observed as a result of the COVID-19 pandemic.(3) For individuals with CCP who are already vulnerable to declining mental health and/or increased substance misuse/abuse, these compounded stresses in combination with decreased mental health-related resources are especially troubling and possibly deadly. Indeed, in our chronic pain clinics the investigators have observed first-hand an increase in the suffering that these patients are enduring since the start of the COVID-19 pandemic including significant increases in the number of early refills of opioid medications, suicides and requests for medical assistance in dying. There is an urgent need to address the mental health and substance use needs of individuals with CCP who have been negatively impacted by the current COVID-19 pandemic.

Transformation in Care Delivery Due To COVID-19 The COVID-19 pandemic has thrust change into the clinical world; telemedicine has become the requisite platform to provide evidence-based solutions addressing the needs of individuals living with chronic pain and struggling with opioid use/misuse during the COVID-19 pandemic.(5,6) Multidisciplinary pain clinics have rapidly adapted and begun to integrate virtual approaches to chronic pain and addiction care across the country;(3,7) however, to our knowledge, none specifically address the unique mental health and substance use needs of individuals with CCP.

The investigators have recently undertaken three innovations to increase accessibility, reach, and efficiency of psychological services within our clinics (GoodHope Ehlers Danlos Syndrome [EDS] Program and the Transitional Pain Service [TPS], both at the Toronto General Hospital [TGH]) that can be leveraged and expanded to address the mental health and substance use needs of patients with CCP within and beyond our clinic at this critical time of need. The first is integration of a mobile app-based pain management solution, Manage My Pain (MMP), into patient care through an established partnership with ManagingLife (the creators of MMP).(8,9) MMP is a patient-driven mobile health solution that aids patients in tracking their symptoms, facilitates communication with providers, and also administers and scores self-report measures. The second innovation is adaptation of existing evidence-based programs into virtual formats, delivered through Ontario Telemedicine Network (OTN), for patients with poor mental health and/or at risk of substance abuse. Of particular interest, the imvestigators developed and piloted a brief, CCP-specific acceptance and commitment therapy (ACT) workshop as this modern, evidence-based form of cognitive-behavioral therapy (CBT) is associated with improved pain acceptance and functioning,(10) significant reductions in depression and anxiety (medium effect size),(11) and decreased opioid use.(12) Even when distilled into a one-visit workshop, ACT is effective in reducing distress, improving functioning and health behaviors, and decreasing opioid use in at-risk medical populations.(12) Internet-based delivery of psychological interventions improves mood in patients with chronic pain,(13) and at least one study has found that online ACT improved mood up to 3 months post-intervention in patients with chronic pain.(14) The third innovation is development of a stepped-care approach to psychological service referral which uses a measurement-based approach to increase efficiency and reduce patient care costs.(15,16) Briefly, this approach consists of screening for mental health concerns (Step 0) followed by offering a one-time ACT workshop to patients who report mental health concerns (Step 1) and, finally, referral to more intensive group programming based in Dialectic Behavior Therapy (DBT) for patients with continued need (Step 2).

This program is well-positioned to make an immediate and important contribution to mental health care for individuals with chronic pain. However, empirical evaluation of this program is still needed. The investigators propose to undertake a prospective, observational study to evaluate the impact and implementation of the virtually-delivered, stepped care mental health program.

Purpose and Objectives The goal this study is to evaluate a newly developed, remote method of identifying individuals with CCP who are at increased risk of poor mental health and/or substance use and provide them with accessible mental health-promoting and substance use-reducing resources during the current COVID pandemic and beyond.

Objectives

1. Investigate the impact of a stepped care mental health program on mental health and substance use risk factors for individuals with chronic pain
2. Examine rates of mental health and substance use risk factors in TPS and EDS clinic patient populations.
3. Examine uptake of the stepped care treatment model amongst patients in the TPS and EDS clinics.

Research Questions:

Can a virtually-delivered stepped care mental health program benefit individuals with complex chronic pain and increased risk for mental health and substance use?

What are current rates of mental health and substance use concerns during the COVID-19 pandemic for individuals in the TPS and EDS clinics?

Will patients in the TPS and EDS clinics participate in a remote mental health and substance use screening and treatment program?

Study Design The investigators propose a prospective, observational study to evaluate the implementation of a remotely-delivered, stepped-care model of psychological treatment. Patients from the GoodHope Ehlers Danlos Syndrome Program and Transitional Pain Service will be invited to complete mental health screening and engage with the self-management application Manage My Pain (Step 0) and, as needed, participate in a one-time Acceptance and Commitment Therapy (Step 1), and a 6-week Dialectic Behavior Therapy Group (Step 2). Patients will be asked to complete self-report measures one-month after participation in each step of the program.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80

Exclusion Criteria:

* Limited comprehension of English
* Known history of serious mental illness (e.g., schizophrenia, dissociative identity disorder)
* Cognitive deficits due to dementia that may affect comprehension (and thereby may limit benefit of the intervention)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients currently being followed by the GoodHope Ehlers Danlos Syndrome Program or the Transitional Pain Service at Toronto General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Medication Misuse | Baseline to post-intervention (3.5 months)
  Measured using the Opioid Risk Tool (ORT). The ORT is a brief self-report tool for assessing risk for opioid misuse/abuse. Patients are asked to acknowledge (yes/no) the presence of Opioid Use risk factors, including family history of substance use, personal history of substance use, age between 16-45, history of preadolescent sexual abuse, and current psychological disorder. Each item is assigned a point value, which differs by respondent gender, and the points for each affirmative response are summed to create a total score. A score of 9 or above has been validated as a marker for increased risk for opioid use disorder for individuals with chronic pain on opioid therapy
Change in Pain Catastrophizing | Baseline to post-intervention (3.5 months)
  Measured using the Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report scale that measures a negative cognitive orientation toward pain, featuring helplessness, magnification, and rumination. Patients are asked to rate the degree to which each statement applies to them on a scale from 0, never, to 4, all the time. A total score of 24 or above has been validated as clinical cut off indicating increased risk of negative pain-related outcomes, mental health issues, and opioid misuse/abuse for individuals with chronic pain.
Change in Depression | Baseline to post-intervention (3.5 months)
  Measured using the Patient Health Questionnaire - 9 (PHQ-9). The PHQ-9 is a 9-item scale designed to capture symptoms of major depressive disorder. Respondents are asked to rate the frequency at which they experience 9 symptoms of depression (e.g. "little interest or pleasure in doing things", "feeling down, depressed, or hopeless") over the past two weeks on a scale from 0, not at all, to 3, nearly every day. Items are summed to create a total score. Clinical cut offs of 5 (mild depression), 10 (moderate depression), and 15 (severe depression) have been determined and validated. The PHQ-9 has been extensively validated for use with chronic pain patients and has also been identified as a risk factor for opioid misuse in this population.
Change in Anxiety | Baseline to post-intervention (3.5 months)
  Measured using the Generalized Anxiety Disorder - 7 (GAD-7). The GAD-7 is a 7-item self-report measure of generalized anxiety. Patients are asked to rate the frequency at which they experience 7 symptoms of generalized anxiety (e.g. "feeling nervous, anxious, or on edge", "not being able to stop or control worrying") over the past two weeks on a scale from 0, not at all, to 3, nearly every day. Clinical cut offs of 5 (mild anxiety), 10 (moderate anxiety), and 15 (severe anxiety) have been determined and validated. This scale has previously been validated as a measure of anxiety symptoms for individuals with chronic pain.
Change in Suicidal Behaviour | Baseline to post-intervention (3.5 months)
  Measured using the Suicide Behaviour Questionnaire - Revised (SBQ-R). The SBQ-R is a 4-item self-report measure of suicide risk. Patients are asked about past suicidal behaviour, current suicidal ideation, communication of suicidal ideation, and perceived likelihood of a future suicide attempt. Responses are summed to create a total score ranging from 3-18. A clinical cut-off of 11 has been recommended as a marker of increased suicide risk.

SECONDARY OUTCOMES:
Change in Pain Intensity | Baseline to post-intervention (3.5 months)
  Pain Numerical Rating Scales
Uptake of the Stepped Care Mental Health Treatment Program | March 2021 to August 2021
  Percentage of those who screen positive that attend a session
Change in Pain Interference | Baseline to post-intervention (3.5 months)
  Measured using the PROMIS Pain Interference Scale 8a. The PROMIS Pain Interference Scale 8a is an eight item self-report measure of pain interference in physical, mental, and social health. Patients are asked to rate the extent to which pain interferes in activities on a scale from 0, not at all, to 5, very much. Responses can be summed to create a total score or compared. The PROMIS pain interference measure has been validated for use as a measure of functioning for individuals with chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hance Clarke, MD, PhD, Principal Investigator — Toronto General Hospital
Locations (1):
- University Health Network- Toronto General Hospital, Toronto, Ontario, Canada